CLINICAL TRIAL: NCT04827810
Title: PH-139: A Phase I Safety and Pharmacokinetic Study of Gamitrinib Administered Intravenously to Patients With Advanced Cancer
Brief Title: A Phase I Safety and Pharmacokinetic Study of Gamitrinib Administered Intravenously to Patients With Advanced Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 21-1045; 1R01CA225913-01A1 (NIH)
Record Dates: First submitted 2021-03-29; First posted 2021-04-01 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Lymphoma; Advanced Solid Tumor
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Dose -1 (Experimental): Accelerated Phase: - Standard Phase: 5 mg
  Interventions: Drug: Gamitrinib
- Dose 1 (Experimental): Accelerated Phase: 10 mg Standard Phase: 10 mg
  Interventions: Drug: Gamitrinib
- Dose 2 (Experimental): Accelerated Phase: 20 mg Standard Phase: 20 mg
  Interventions: Drug: Gamitrinib
- Dose 3 (Experimental): Accelerated Phase: 40 mg Standard Phase: 35 mg
  Interventions: Drug: Gamitrinib
- Dose 4 (Experimental): Accelerated Phase: 80 mg Standard Phase: 50 mg
  Interventions: Drug: Gamitrinib
- Dose 5 (Experimental): Accelerated Phase: 160 mg Standard Phase: 65 mg
  Interventions: Drug: Gamitrinib
- Dose 6 (Experimental): Accelerated Phase: 320 mg Standard Phase: 85 mg
  Interventions: Drug: Gamitrinib

INTERVENTIONS:
Drug: Gamitrinib — This is a first-in-human, phase I, open-label, non-randomized dose-escalation and dose-expansion study with the primary objective to determine the safety profile of small molecule, mitochondrial-targeted Hsp90 inhibitor, gamitrinib, including identification of dose-limiting toxicities (DLT) and maximum tolerated dose (MTD) in patients with advanced cancers. A secondary objective of the study is to determine the recommended dose and regimen(s) for a phase II study. This study is based on preclinical data demonstrating the anticancer activity, unique mechanism of action and preliminary safety of gamitrinib.

SUMMARY:
This is a first-in-human, phase I, open-label, non-randomized dose-escalation and dose-expansion study with the primary objective to determine the safety profile of small molecule, mitochondrial-targeted Hsp90 inhibitor, gamitrinib, including identification of dose-limiting toxicities (DLT) and maximum tolerated dose (MTD) in patients with advanced cancers. A secondary objective of the study is to determine the recommended dose and regimen(s) for a phase II study. This study is based on preclinical data demonstrating the anticancer activity, unique mechanism of action and preliminary safety of gamitrinib.

In the dose-finding portion of this study, gamitrinib formulated in Lipoid S100®-based formulation will be administered as a 1-hour IV infusion once weekly for four weeks as 28-day treatment cycles. Up to 36 patients will be enrolled in the dose-escalation component of the study based on anticipated cohorts. The starting dose will be 10 mg, corresponding to allometric scaling) from the most sensitive species (rats) in the 29-day GLP toxicology and toxicokinetic studies with 14-day recovery period of gamitrinib. Dose-escalation will follow a 3+3 design. Six patients will be enrolled in the dose-expansion component of the study at MTD for the purpose of exploring pharmacodynamic effects via tumor pre and on-therapy biopsies.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of advanced cancer refractory to standard of care therapy, or for whom no standard of care therapy is available. Any numbers of prior therapies are allowed.
* Dose escalation phase: Solid tumors and lymphoma may have measurable or evaluable disease as per Response Evaluation Criteria in Solid Tumors (RECIST v. 1.1) or as per RECIL 2017 criteria
* Dose expansion phase:

  i. All patients must have at least one site of measurable disease as defined by RECIST v. 1.1. or RECIL 2017, for solid tumors and lymphoma, respectively ii. Patients in the expansion cohort must have at least one non-target lesion deemed safe to biopsy, in the opinion of the investigator, and be willing to undergo mandatory core biopsies. This includes pre-treatment and an on-treatment biopsy. Biopsies at the time of progression are highly desired, but optional.

iii. The lesion(s) which will be used for response assessment may not be biopsied iv. Target lesions that have been previously irradiated will not be considered measurable unless increase in size is observed following completion of radiation therapy

* All previous therapies of cancer, including radiotherapy major surgery and investigational therapies must be discontinued for ≥14 days (≥ 28 days for mitomycin C or nitrosoureas) before Cycle 1 Day 1 (C1D1), and all acute effects of any prior therapy must have resolved to baseline severity or Grade ≤ 1 Common Terminology Criteria for Adverse Events (CTCAE v5), except alopecia or parameters defined in this eligibility list.
* Age > 18 years.
* ECOG performance status 0- 2
* Patients must have normal organ and marrow function as defined below
* Absolute neutrophil count ≥1,500/mm3 without growth factor use ≤ 7 days prior to C1D1 Platelets ≥85,000/mm3 without platelet transfusion ≤ 7 days prior to C1D1 Hemoglobin >8.5 mg/dL without red blood cell transfusion ≤ 7 days prior to C1D1 Total serum bilirubin <1.5 X upper limit of normal (ULN) (except for patients with documented Gilbert's syndrome) AST (SGOT)/ALT (SGPT) ≤2 X ULN; ≤ 5 X ULN if liver dysfunction is felt to be secondary to tumor burden Serum creatinine ≤ 1.5 X ULN (OR creatinine clearance ≥ 60 mL/min/1.73 m2) Serum or urine pregnancy test (WOCBP only) negative ≤7 days of C1D1
* Ability to understand and willingness to sign a written informed consent, HIPAA consent document and comply with the study scheduled visits, treatment plans, laboratory tests and other procedures.
* Female patients must be surgically sterile or be postmenopausal, or must agree to use effective contraception during the period of the trial and for at least 90 days after completion of treatment. Male patients must be surgically sterile or must agree to use effective contraception during the period of the trial and for at least 90 days after completion of treatment. The decision of effective contraception will be based on the judgment of the principal investigator or a designated associate.

Exclusion Criteria:

* Patients with symptomatic brain metastases are excluded. Patients with asymptomatic and treated CNS metastases may participate in this trial. The patient must have completed any prior treatment for CNS metastases > 28 days prior to study entry, including radiotherapy or surgery. Concurrent use of steroids for the treatment of brain metastasis are not permitted.
* Current treatment on another (therapeutic) clinical trial
* Hypertension not adequately controlled with medications (>150/100 mm Hg despite optimal medical therapy)
* Active bacterial fungal or viral infection including hepatitis B (HBV), hepatitis C (HCV), requiring treatment with IV antibiotic, IV anti-fungal, or anti-viral (Testing is not required for eligibility).
* Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness (testing is not required for eligibility).
* Any of the following in the previous 6 months: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident, transient ischemic attack or symptomatic pulmonary embolism.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, or in the judgment of the investigator would make the patient inappropriate for entry into the study
* Pregnant or breast feeding. Refer to section 4.4 for further detail.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2021-11-05 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Determine the MTD and/or RP2D of gamitrinib when administered once weekly. | 7 years
  First cycle dose-limiting toxicities. The maximally tolerated dose (MTD) is defined as the dose level below which the absolute observed DLT rate is > 25%. The MTD is equivalent to the anticipated recommended phase 2 dose (RP2D).

SECONDARY OUTCOMES:
Evaluate the overall safety profile of intravenously administered single-agent gamitrinib | 7 years
  Overall, safety profile of gamitrinib as characterized by type, frequency, severity, timing and relationship to study therapy of adverse events and laboratory abnormalities according to NCI CTCAE v5.0.
To evaluate the peak concentration (Cmax) of gamitrinib | 7 years
  Blood sample will be collected for determination of gamitrinib plasma concentrations. The PK parameter to be evaluated includes peak concentration (Cmax).
To evaluate the area under the concentration time curve (AUC0-t) of gamitrinib | 7 years
  Blood sample will be collected for determination of gamitrinib plasma concentrations. PK parameter to be evaluated includes area under the concentration time curve (AUC0-t).
To evaluate the clearance (CL) of gamitrinib | 7 years
  Blood sample will be collected for determination of gamitrinib plasma concentrations. PK parameter to be evaluated includes clearance (CL).
To evaluate the time to maximum concentration (Tmax) of gamitrinib | 7 years
  Blood sample will be collected for determination of gamitrinib plasma concentrations. PK parameter to be evaluated includes time to maximum concentration (Tmax).
To evaluate the coefficient of variation (CV) of gamitrinib | 7 years
  Blood sample will be collected for determination of gamitrinib plasma concentrations. A coefficient of variation (CV) will be assessed at each dose level.
Assess the pharmacodynamic effects of gamitrinib | 7 years
  Assessment of gamitrinib effects on pharmacodynamic markers. The processed samples will be profiled for changes in the expression of 301 metabolites by Ultrahigh Performance Liquid Chromatography/Mass Spectrometry (UPLC/MS) or Gas Chromatography/Mass Spectrometry (G/MS) using the Metabolon, Inc. discovery platform
Document any anti-tumor activity of single agent gamitrinib | 7 years
  Objective tumor response, as assessed using RECIST 1.1 and RECIL 2017 criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hayat U, Elliott GT, Olszanski AJ, Altieri DC. Feasibility and safety of targeting mitochondria for cancer therapy - preclinical characterization of gamitrinib, a first-in-class, mitochondriaL-targeted small molecule Hsp90 inhibitor. Cancer Biol Ther. 2022 Dec 31;23(1):117-126. doi: 10.1080/15384047.2022.2029132. PMID 35129069